CLINICAL TRIAL: NCT04010162
Title: Social Media Awareness Level of Non-urogynecologist Doctors About the Current Mesh Discussions in Urogynecology: A Practical Survey Study.
Brief Title: Mesh Debate Awareness Among Non-urogynecologists. A Practical Survey Study.
Acronym: Mesh_Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Adnan Orhan, Medical Doctor, Researcher, Obstetrician and Gynecologist, Uludag University
Other Study IDs: UU-SUAM-MREC-2018-13/11
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence; Complication of Surgical Procedure
Keywords: mesh complications; social media awareness; knowledge of doctors
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group-1: King's College Hospital: Doctors in King's College Hospital, London, The United Kingdom (Excluding Urology and Gynecology)
  Interventions: Other: Mesh debate awareness survey
- Group-2: Uludag University Hospital: Doctors in Uludag University Hospital, Bursa, Turkey (Excluding Urology and Gynecology)
  Interventions: Other: Mesh debate awareness survey
- Group-3: The United States: Doctors from The United States (Excluding Urology and Gynecology)
  Interventions: Other: Mesh debate awareness survey
- Group-4: The World: Doctors from all over the world (Excluding Urology and Gynecology)
  Interventions: Other: Mesh debate awareness survey

INTERVENTIONS:
Other: Mesh debate awareness survey — A web-based questionnaire with questions about recent discussions of mesh in urogynecology.
  10 questions. Average survey completion time: 1 minute

SUMMARY:
This study evaluates the awareness of mesh discussions in urogynecology among non-urogynecologists. A web-based questionnaire will be sent to four groups. Group-1 is King's College Hospital doctors. Group-2 is Uludag University Hospital doctors. Group-3 is doctors from the United States, and Group-4 is doctors from all over the world.

DETAILED DESCRIPTION:
There has been a great deal of discussion about mesh complications in urogynecology. During the following decade, vaginal mesh operations for pelvic organ prolapse increased exponentially all over the world, particularly in the United States. Once the complications started to increase, the publication of mesh-related complications on social and broadcast media and the increase of medico-legal claims the United States led to an extensive FDA (Food and Drug Administration) restriction on vaginal mesh procedures in 2013. On January 5, 2016, the FDA reclassified surgical mesh for transvaginal repair of the pelvic organ prolapse into class III, which require premarket approval. Finally, on April 16, 2019, the FDA ordered all manufacturers of urogynecological mesh intended for transvaginal repair to stop selling and distributing their products immediately. However, awareness of the other doctors in branches of medicine outside of gynecology and urology is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Doctors from all branches of medicine
* Basic sciences: Immunology, Medical Biochemistry, Microbiology and Infectious Diseases, Forensic Medicine, Family Medicine, Public Health, Medical genetics, Medical pharmacology.
* Pediatrics: Pediatric allergy, Pediatric respiratory, Pediatric dentistry, Pediatric endocrinology, Pediatric gastroenterology and nutrition, Pediatric haematology, Pediatric nephrology, Pediatric neurology, Pediatric oncology, Pediatric ophthalmology, Pediatric surgery, Child and adolescent psychiatry, Pediatric orthopedics.
* Basic internal medicine specialties: Gastroenterology, Medical Oncology, Rheumatology, Hematology, Nephrology, Endocrinology
* Other internal medicine specialties: Neurology, Nuclear medicine, Radiology, Radiation Oncology, Psychiatry, Sport medicine, Respiratory medicine, Physical medicine and rehabilitation, Geriatrics, Dermatology, Cardiology
* Surgical Departments: Emergency and Accident Medicine, Heart and vascular surgery, Ophthalmatology, Orthopedics and Traumatology, Plastic and reconstructive surgery, Medical pathology, Anesthesiology and reanimation, Neurosurgery, General surgery, Chest surgery

Exclusion Criteria:

* Obstetricians and Gynaecologists,
* Urogynecologists,
* Urologists,
* Perinatologists ,
* Gynecological Oncologists,
* Doctors from Reproductive Endocrinology and Infertility,
* Uro-oncologists
* Andrologists.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Doctors from four different groups (1-KCH, 2-UUH, 3-USA, 4-WORLD) are expected to complete the questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
Awareness of the current mesh discussion in urogynecology. | 1 minute
  Web-based survey about current mesh discussion in Urogynecology with ten simple questions will be answered by the doctors in four groups (Question-8).

SECONDARY OUTCOMES:
Social media awareness about the mesh discussions in urogynecology | 1 minute
  Web-based survey about current mesh discussion in Urogynecology with ten simple questions will be answered by the doctors in four groups (Question-10).

CONTACTS AND LOCATIONS:
Overall Officials: Kemal Ozerkan, M.D., Study Director — Uludag University
Locations (1):
- Uludag University Hospital, Department of Obstetrics and Gynecology, Bursa, Ozluce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lensen EJ, Withagen MI, Kluivers KB, Milani AL, Vierhout ME. Surgical treatment of pelvic organ prolapse: a historical review with emphasis on the anterior compartment. Int Urogynecol J. 2013 Oct;24(10):1593-602. doi: 10.1007/s00192-013-2074-2. Epub 2013 Mar 15. PMID 23494056
- [Background] LANE FE. Repair of posthysterectomy vaginal-vault prolapse. Obstet Gynecol. 1962 Jul;20:72-7. doi: 10.1097/00006250-196207000-00009. No abstract available. PMID 14462011
- [Background] Maher C, Feiner B, Baessler K, Christmann-Schmid C, Haya N, Brown J. Surgery for women with anterior compartment prolapse. Cochrane Database Syst Rev. 2016 Nov 30;11(11):CD004014. doi: 10.1002/14651858.CD004014.pub6. PMID 27901278
- [Background] Nygaard IE, McCreery R, Brubaker L, Connolly A, Cundiff G, Weber AM, Zyczynski H; Pelvic Floor Disorders Network. Abdominal sacrocolpopexy: a comprehensive review. Obstet Gynecol. 2004 Oct;104(4):805-23. doi: 10.1097/01.AOG.0000139514.90897.07. PMID 15458906